CLINICAL TRIAL: NCT01153737
Title: Primary Care Randomized Clinical Trial: Manual Therapy Effectiveness in Comparison With TENS in Patients With Neck Pain
Brief Title: Manual Therapy Effectiveness in Comparison With Electric Nerve Stimulation (TENS) in Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia Atencion Primaria Area 3 (Other Government)
Collaborators: University of Alcala (Other)
Responsible Party: Esperanza Escortell, Gerencia Atencion Primaria Area 3
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04/1320
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Neck Pain
Keywords: Neck pain; Primary Health Care; Manual Therapy; TENS
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- manual therapy (Experimental)
  Interventions: Other: Manual therapy (MT)
- TENS (Active Comparator): Electric Nerve Stimulation (TENS)
  Interventions: Other: TENS

INTERVENTIONS:
Other: Manual therapy (MT) — Ten treatment sessions of 30 minutes of MT or TENS on alternate days were provided by primary care physical therapists. MT techniques: neuromuscular technique, postisometric stretching, spray and stretching and Jones technique.
  Arms: manual therapy
Other: TENS — Ten treatment sessions of 30 minutes of MT or TENS on alternate days were provided by primary care physical therapists. TENS electrode placement were: in the painful area, in the metamere or in the nerve´s pathway. It was applied at a frequency of 80 Hz, with ≤150 µs pulse duration and adjusted amplitude.
  Arms: TENS

SUMMARY:
This study investigated effectiveness of manual therapy (MT) with Electric Nerve Stimulation (TENS) to reduce pain intensity in patients with mechanical neck disorder (MND). A randomized multi-centered controlled clinical trial was performed in 12 Primary Care Physiotherapy Units in Madrid Region.

DETAILED DESCRIPTION:
The purpose of tis study is to evaluate the effectiveness of manual therapy (MT) with Electric Nerve Stimulation (TENS) to reduce pain intensity in patients with mechanical neck disorder (MND). Design: randomized multi-centered controlled clinical trial. Location: 12 Primary Care Physiotherapy Units in Madrid Region. Ninety patients were included with diagnoses of subacute or chronic MND without neurological damage, 47 patients received MT and 43 TENS. The primary outcome was pain intensity measured in millimeters using the Visual Analogue Scale. Also disability, quality of life, adverse effects and sociodemographic and prognosis variables were measured. Three evaluations were performed (before, when the procedure finished and six months after). Seventy one patients (79%) completed the follow-up measurement at six months. In more than half of the treated patients the procedure had a clinically relevant "short term" result after having ended the intervention, when either MT or TENS was used. The success rate decreased to one third of the patients 6 months after the intervention. No differences can be found in the reduction of pain, in the decrease of disability nor in the quality of life between both therapies. Both analyzed physiotherapy techniques produce a short term pain reduction that is clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* diagnoses of subacute or chronic MND without neurological damage, according to the Classification of the Quebec Task Force on Spinal Disorders (Spitzer 1987);
* full physical and psychological capacity to follow the clinical trial's requirements;
* consent to participate

Exclusion Criteria:

* Signs of neurological damage according to the Neurologic Screening Checklist (Hoving et al. 2002),
* pregnant women,
* previous neck rachis surgery,
* patients who received physical therapy or an alternative treatment of the neck or shoulder 6 months prior to the beginning of the study,
* patients who intended to receive other treatments during the study
* patients with important psychiatric disorders or other health problems that would contraindicate the techniques to be used (i.e. pacemaker).
* Patients with neck pain caused by an inflammatory, neurological or rheumatic disease, severe osteoporosis, fracture, luxation or vertebrobasilar insufficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured in millimeters (Visual Visual Analogue Scale, VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Esperazna Escortell, MD, Principal Investigator — Servicio Madrileño de Salud, Madrid, Spain
Locations (1):
- Servicio Madrileño de Salud, Madrid, Spain

REFERENCES:
- [Background] Escortell Mayor E, Lebrijo Perez G, Perez Martin Y, Asunsolo del Barco A, Riesgo Fuertes R, Saa Requejo C; TEMA-TENS Group. [Randomized clinical trial for primary care patients with neck pain: manual therapy versus electrical stimulation]. Aten Primaria. 2008 Jul;40(7):337-43. doi: 10.1157/13124126. Spanish. PMID 18620635
- [Background] Escortell-Mayor E, Riesgo-Fuertes R, Garrido-Elustondo S, Asunsolo-Del Barco A, Diaz-Pulido B, Blanco-Diaz M, Bejerano-Alvarez E; TEMA-TENS Group. Primary care randomized clinical trial: manual therapy effectiveness in comparison with TENS in patients with neck pain. Man Ther. 2011 Feb;16(1):66-73. doi: 10.1016/j.math.2010.07.003. Epub 2010 Aug 5. PMID 20691631
- [Background] Elustondo SG, Fuertes RR, Mayor EE, del Barco AA, Martin YP, Castro BM. Satisfaction of patients with mechanical neck disorders attended to by primary care physical therapists. J Eval Clin Pract. 2010 Jun;16(3):445-50. doi: 10.1111/j.1365-2753.2009.01138.x. Epub 2010 Mar 10. PMID 20337831
- [Result] Escortell Mayor E, Lebrijo Perez G, Sanchez Sanchez B, Asunsolo del Barco A. [Difficulties in carrying out public projects of investigation in primary care]. Aten Primaria. 2008 Oct;40(10):536-7. doi: 10.1157/13127242. No abstract available. Spanish. PMID 19054468